CLINICAL TRIAL: NCT06801938
Title: Comparison of Complications Detected by Perioperative Cystoscopy Combined With Methylene Blue Test and Postoperative Cystoscopy in TVT and TOT Operations
Brief Title: Evaluation of Perioperative Cystoscopy and Methylene Blue Test in Detecting Complications in TVT and TOT Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GaziosmanpasaTREHfkgfkg
Record Dates: First submitted 2025-01-25; First posted 2025-01-30 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Incontinence Stress
Keywords: tvt; tot; cystoscopy
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: The ability of perioperative methylene blue test and postoperative cystoscopy to detect complications in patients with stress urinary incontinence will be compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perioperative Methylene Blue and Cystoscopy with Postoperative Cystoscopy for Complication Detection (Experimental): This arm includes patients with stress urinary incontinence who will undergo perioperative methylene blue test and cystoscopy, followed by postoperative cystoscopy to detect any complications. The aim is to assess the ability of these methods to identify complications in the postoperative period.
  Interventions: Procedure: Perioperative Cystoscopy and Methylene Blue Test

INTERVENTIONS:
Procedure: Perioperative Cystoscopy and Methylene Blue Test — The ability of perioperative methylene blue and cystoscopy versus postoperative cystoscopy to detect complications will be compared in patients.
  Other Names: postoperative cystoscopy

SUMMARY:
Comparison of complications detected by perioperative cystoscopy combined with methylene blue test and postoperative cystoscopy in TVT and TOT operations.

ELIGIBILITY:
Inclusion Criteria:

* Providing consent to participate in the study
* Being between the ages of 18 and 85
* Having stress urinary incontinence
* No active cardiac disease
* No connective tissue disorders (e.g., Marfan syndrome)
* No known gynecological malignancy
* BMI under 30
* No chronic constipation
* No inflammatory bowel disease

Exclusion Criteria:

* Not providing consent to participate in the study
* Being under 18 or over 85 years old
* Not having stress urinary incontinence
* Having active cardiac disease
* Having connective tissue disorders (e.g., Marfan syndrome)
* Having a known gynecological malignancy
* Having a BMI over 30
* Having chronic constipation
* Having inflammatory bowel disease

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
rate of complication detection | 6 months
  Specifically, it would compare the ability of the perioperative methylene blue test and cystoscopy versus postoperative cystoscopy to detect complications. This measure will be used to evaluate the accuracy and effectiveness of both methods

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpaşa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No